CLINICAL TRIAL: NCT01798654
Title: Safety of Endoscopic Ultrasound-guided Fine Needle Aspiration for Patients With Antithrombotic Agents
Brief Title: EUS-FNA for Patients With Antithrombotic Agents
Status: Completed | Type: Observational
Sponsor: Hokkaido Pancreatobiliary Endoscopic Intervention Study Group (Network)
Collaborators: Hokkaido University Hospital (Other)
Responsible Party: Principal Investigator, Kazumichi Kawakubo, M.D. and Ph.D., Hokkaido Pancreatobiliary Endoscopic Intervention Study Group
Other Study IDs: H-Spirit1201
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Antithrombotic agents

SUMMARY:
The purpose of this study to evaluate a safety of endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) for patients with antithrombotic agents.

ELIGIBILITY:
Inclusion Criteria:

* Undergo EUS-FNA
* take antithrombotic agents

Exclusion Criteria:

* Cystic lesion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In hospital
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Patients who suffered bleeding complication | One week

CONTACTS AND LOCATIONS:
Locations (1):
- Hokkaido University Graduate School of Medicine, Sapporo, Japan